CLINICAL TRIAL: NCT00647205
Title: Evaluation of 2 Interferon γ Assays (QuantiFERON TB Gold In-Tube® and T-SPOT.TB®) in the Diagnosis of Latent Tuberculosis in HIV-infected Patients.ANRS EP 40 QUANTI SPOT
Brief Title: Evaluation of 2 Interferon γ Assays in the Diagnosis of Latent Tuberculosis in HIV-infected Patients.ANRS EP 40 QUANTI SPOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Marcia Trumeau regulatory, ANRS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ANRS EP 40 QUANTI SPOT
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Interferon, gamma; HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Sham Comparator): HIV infected antiretroviral naïve patients originated from low TB prevalence countries without any active TB with CD4 cell count > 350/mm3
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®
- 2 (Sham Comparator): HIV infected antiretroviral naïve patients originated from low TB prevalence countries without any active T with CD4 < 350/mm3)
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®
- 3 (Sham Comparator): HIV infected antiretroviral naïve patients originated from high TB prevalence countries without any active TB with CD4 < 350/mm3)
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®
- 4 (Sham Comparator): HIV infected antiretroviral naïve patients originated from high TB prevalence countries without any active TB with CD4 > 350/mm3)
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®
- 5 (Sham Comparator): HIV infected patients with active TB
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®
- 6 (Sham Comparator): HIV negative patients with active TB
  Interventions: Device: QuantiFERON TB Gold In-Tube; Device: T-SPOT.TB®

INTERVENTIONS:
Device: QuantiFERON TB Gold In-Tube
Device: T-SPOT.TB®

SUMMARY:
The aim of this study is to estimate the usefulness of QuantiFERON TB Gold In-Tube® and T-SPOT.TB® for the diagnosis of latent tuberculosis in HIV infected antiretroviral naive patients: 80 originated from low TB prevalence countries, without any active TB; 80 HIV infected antiretroviral naïve patients originated from high TB prevalence countries, without any active TB, 40 HIV infected patients with active TB and 40 HIV negative patients with active TB.

DETAILED DESCRIPTION:
The aim of this study is to estimate the usefulness of QuantiFERON TB Gold In-Tube and T-SPOT.TB for the diagnosis of latent tuberculosis in this population. Concordance between TST, QuantiFERON TB Gold and T-SPOT.TB will be assessed in patients with different risks of TB, in a transversal study. This study will include 240 patients during 2 years: 80 HIV infected antiretroviral naïve patients originated from low TB prevalence countries, without any active TB (40 patients with CD4 cell count > 350/mm3, 40 with CD4 < 350/mm3), 80 HIV infected antiretroviral naïve patients originated from high TB prevalence countries, without any active TB, 40 HIV infected patients with active TB and 40 HIV negative patients with active TB. TST and the 2 blood interferon gamma assay will be compared according to the level of risk. The improvement of latent TB diagnosis in HIV infected patients may lead to the initiation of TB prophylaxis and decrease the incidence of this life threatening disease.

ELIGIBILITY:
Inclusion Criteria:

* sign an informed consent
* to be adult
* not to be pregnant
* to have a clinical examination and a medical questionnaire

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Intradermal Tuberculin Tests QuantiFERON TB Gold In-Tube® T-SPOT.TB® | 48 to 72 hours after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bonnet, MD, Principal Investigator — AP-HP Paris; France Mentre, PHD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service des Maladies Infectieuses B Hopital Bichat, Paris, France